CLINICAL TRIAL: NCT05553951
Title: Adherence in Global Airways - Difference Between Structured and Systematic Nursing Supervison vs Usual Care
Brief Title: Adherence in Global Airways
Acronym: AIR2022
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Christiane Haase (Other)
Responsible Party: Sponsor-Investigator, Christiane Haase, Clinical nurse specialist and Phd-student, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-ENT-2- adherence
Record Dates: First submitted 2022-09-14; First posted 2022-09-26 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Chronic Rhinosinusitis Without Nasal Polyps; Asthma; Chronic Rhinosinusitis With Nasal Polyps; Chronic Rhinosinusitis (Diagnosis)
Keywords: Adherence; Nurse; Global airways; Astma; Chronic Rhinosinusitis with Nasal Polyps
MeSH Terms: conditions — Asthma; Disease | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventions group (Experimental): will receive systematic and structured nursing supervison about their adherence
  Interventions: Behavioral: Intervention
- Control group (Placebo Comparator): Will receive usual care
  Interventions: Behavioral: Controlgroup

INTERVENTIONS:
Behavioral: Controlgroup — The control group and intervention group will receive daily text message reminders twice a week to take their medications and to rinse their nose.
  Arms: Control group
Behavioral: Intervention — Patients in the intervention group will receive systematic and structured nursing guidance regarding their adherence, which includes proper use of nasal irrigation once or twice daily, nasal steroid/drops, use of inhaled medications, follow-up of smoking status. The intervention group will receive guidance videos which have been prepared prior to the study and will be standard for the intervention group. Guidance videos will cover the correct use of nasal irrigation, inhalation steroid, and nasal steroid/drops.
  Arms: Interventions group

SUMMARY:
There is a strong case for treating diseases of both the upper and lower airways (global airways) simultaneously because they share the same inflammatory mechanisms. About 9% have chronic sinusitis (CRS) and 4% of the Danish population are diagnosed with CRS with nasal polyps (CRSwNP)) and 7-10% have asthma. CRS has a multifactorial background, with CRSwNP characterized by Type 2 inflammation, and approximately 50% with Type 2 CRSwNP also have co-morbid asthma. Well-treated CRS has an impact on asthma control, and well-treated asthma has an impact on CRS.

Several studies show that patients with asthma have low adherence, but only a few if any of studies are available on adherence in CRS.

Aim:

To investigate the effect of systematic and structured nursing supervision in patients with CRSwNP and asthma primarily on adherence.

Hypothesis and research questions: Patients with respiratory diseases can improve their adherence to their non-medical and medical treatment for CRSwNP/CRS and asthma by systematic and structured nursing supervision compared to patients who receive usual care.

In a randomized clinical trial, we will investigate whether the level of adherence measured by the questionnaire MARS-5-N and MARS-5- L in patients with CRSwNP and asthma can be improved by 7 points after systematic and structured nursing guidance at baseline visit and controlled after four months - compared with those patients who have not received the above guidance.

Primary outcome: is change in adherence rate measured by the MARS-5-N/L questionnaire in patients with CRSwNP and asthma can be improved by 4 points after systematic and structured nursing guidance at the initial visit and controlled after four months - compared with patients who have not received the above guidance.

Inclusion Criteria:

Adherence to MARS- 5 L/N ≤35 at first visit, diagnosed with asthma (with/without allergic rhinitis) at initial visit, diagnosed with CRSwNP, able to use smartphone, ACQ ≥1.2 or ACT≤15 (partially uncontrolled asthma), >18 years of age, SNOT-22 score ≥35

Exclusion Criteria:

* Adherence to MARS-5- L/N >35 points at first visit,do not have smartphone, does not read/speak English, other illness requiring regular medication, pregnancy/pregnancy that started during the study, server psychological comorbidities

Questionnaires: Patients must answer the following questionnaires at baseline and at 4 months follow up ESS, SNOT-22, ACQ-7, ACT, MiniAqLq, HADS, STARR-15

ELIGIBILITY:
Inclusion Criteria:

* Adherence to MARS- 5 L/N ≤35 at first visit
* Diagnosed with asthma (with and without allergic rhinitis) at initial visit
* Able to use smartphone
* ACQ ≥1.2 or ACT≤15 (partially uncontrolled asthma)
* Be over 18 years of age
* SNOT-22 score ≥35
* Diagnosed with CRSwNP

Exclusion Criteria:

* Adherence to MARS-5- L/N >35 points at first visit
* Do not have smartphone
* Does not read or speak English
* Other illness requiring regular medication
* Pregnancy and pregnancy that started during the study time period
* Servere psychological comorbidities

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
MARS-5 L/N - Medication adherence report scale both for upper and lower airways | 4 months
  Min. 0 point= non adherent, max. 25 point=adherent

SECONDARY OUTCOMES:
SNOT-22 - The Sino-Nasal Outcome Test 22 | 4 months
  min. 0 point=no symptoms, max. 110 point=many symptoms.
miniAQLQ - Mini asthma quality of life questionnaire | 4 months
  min. 1= all the time, max. 7= not at all
HADS - Hospital Anxiety and Depression Scale | 4 months
  Min 0 point=no risk, Max 21 point=high risk. It applies both anxiety and depression
STARR-15 ) Standard test for asthma, rhinitis and chronic rhinosinusitis (15 questions) | 4 months
  There is no minimum or maximum yet
ACT - Asthma Control Test | 4 months
  min. 5 (poor control of asthma), max. 25 (complete control of asthma),
ACQ-7 - Asthma Control Questionnaire | 4 months
  min. 0 point= complete control of asthma, max 6 point= poor control of asthma Rigtig dårlig kontrol er > 1.5
ESS - EPWORTH SLEEPINESS SCALE | 4 months
  min=0 point= normal sleep, max. 24 point= severe sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke P Backer, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Department of Otorhinolaryngology, Head and Neck Surgery & Audiology, Copenhagen, Denmark

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT05553951/Prot_SAP_ICF_000.pdf